CLINICAL TRIAL: NCT01985802
Title: Optimal Pacing in Patients With First-degree AV-block
Brief Title: Pacing in First-degree AV-block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048871
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: First-degree AV-block; Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pacing - Cross-over (Other): Pacing will be conducted in 3 different ways (atrial, dual chamber and His-bundle pacing) at 2 different rates (basal and 100 bpm).
  Interventions: Other: Pacing

INTERVENTIONS:
Other: Pacing
  Other Names: Additional catheter may be used to evaluate heart performance during pacing. Does not require additional IV access

SUMMARY:
The purpose of this study is to explore if there is a less harmful way to pace patients with first-degree AV-block to ensure that the negative effects inferred by the pacing do not outweigh the positive effects of AV-synchrony. The main hypothesis of the study is that His-bundle pacing will offer a more physiological mode of pacing in patients with first-degree AV-block than conventional pacing.

Patients scheduled for catheter ablation of atrial fibrillation (AF) in sinus rhythm, with first degree AV-block, normal QRS duration less than 120 ms and normal left ventricular ejection fraction will be included. During the AF ablation three different pacing modes (atrial, AV-synchronous and His-bundle pacing) at two different rates (5 to10 bpm above the basal rate and at 100 bpm) will be performed and evaluated using echocardiography. After the completion of all six pacing protocols (i.e., three modes at two different rates) the experimental part of the procedure ends.

The primary end-point will be echocardiographic evidence of dyssynchrony. Secondary end-points will include left ventricular ejection fraction, left ventricular volume, mitral regurgitation, septal to posterior wall motion delay and inter-ventricular wall motion delay. Since the research study is conducted in parallel with the standard catheter ablation, we do not anticipate any additional side effects as a result of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for catheter ablation of atrial fibrillation in sinus rhythm and PR prolongation exceeding or equal to 200 ms
* QRS duration less than 120 ms
* Normal left ventricular ejection fraction on echocardiography.

Exclusion Criteria:

* Any bundle branch block
* Second- or third-degree AV-block
* Congestive heart failure, cardiomyopathy, myocardial infarction or major surgical procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Echocardiographic evidence of dyssynchrony (AV, intra- or inter-ventricular) | During each step of the pacing procedure the echocardiographic data will be recorded; over approximately 5-10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: James P Daubert, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States